CLINICAL TRIAL: NCT02373137
Title: Descemet Endothelial Thickness Comparison Trial
Acronym: DETECT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oregon Health and Science University (Other)
Collaborators: University of California, San Francisco (Other); Stanford University (Other)
Responsible Party: Principal Investigator, Winston Chamberlain, MD, PhD, Ophthalmologist, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00010818
Record Dates: First submitted 2015-01-27; First posted 2015-02-26 (Estimated); Results first posted 2019-07-02 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Keratoplasty; Grafting, Corneal; Transplantation, Corneal; Transplantation, Cornea; Keratoplasty, Lamellar
MeSH Terms: conditions — Corneal Diseases | interventions — Prednisolone; Methylprednisolone; Ofloxacin; Tropicamide; Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DSAEK (Other): Type of corneal transplant; Tissue grafts will be cut to the right thickness using a microkeratome prepared at the eye bank per standard eye bank protocol (about 60-90 microns thick). A 4 mm corneal incision will be used, with Endoserter as the means of inserting the graft, an FDA approved device for this purpose.
  Interventions: Procedure: DSAEK; Device: Endoserter; Drug: Prednisolone; Drug: Ofloxacin; Drug: Tropicamide; Drug: Phenylephrine
- DMEK (Other): Type of corneal transplant; Endothelial grafts will be pre-peeled at the eyebank (70%). In the operating room the remaining 30% will be peeled, and the endothelium will be stained with trypan blue. A 3.5 mm corneal incision will be used and the graft will be inserted with a modified jones tube injector. The tap technique will be used to position the graft.
  Interventions: Procedure: DMEK; Drug: Prednisolone; Drug: Ofloxacin; Drug: Tropicamide; Drug: Phenylephrine; Device: Jones Tube

INTERVENTIONS:
Procedure: DSAEK
  Arms: DSAEK
Procedure: DMEK
  Arms: DMEK
Device: Endoserter — The Endoserter, a corneal endothelium device, is an approved FDA device. This will be used to insert and position the graft into the anterior chamber during endothelial replacement surgery. It is a sterile, single-use instrument.
  Arms: DSAEK
Drug: Prednisolone — Prednisolone is a corticosteroid used to alleviate swelling post-surgery.
  Other Names: Millipred; Orapred; Omnipred; Econopred; Flo-Pred
Drug: Ofloxacin — Ofloxacin is an antibiotic used to treat bacterial infections of the eye.
  Other Names: Ocuflox; Floxin
Drug: Tropicamide — Tropicamide is a prescription drug used to dilate pupils during an eye exam.
  Other Names: Mydriacyl
Drug: Phenylephrine — Phenylephrine is a prescription drug used to dilate pupils during an eye exam.
Device: Jones Tube — The Jones Tube will be used to insert the graft into a 3.5 mm corneal incision during endothelial replacement surgery.
  Arms: DMEK

SUMMARY:
The purpose of this study is to compare visual acuity outcomes of two types of endothelial keratoplasty: 1) Ultrathin Descemet's Stripping Endothelial Keratoplasty (DSAEK) or 2) Descemet's Membrane Endothelial Keratoplasty (DMEK). Half of the participants will be randomized to have DSAEK and the other half will have DMEK.

DETAILED DESCRIPTION:
Corneal transplantation has evolved rapidly in recent years. Lamellar keratoplasty to replace diseased endothelium has led to faster recovery times, fewer complications, and better visual acuity outcomes. Currently, Descemet's Stripping Endothelial Keratoplasty (DSAEK) is the most common procedure because of its relative ease and good outcomes. Newer techniques such as Descemet's Membrane Endothelial Keratoplasty (DMEK), where Descemet's membrane alone is transplanted, has the potential to further improve visual acuity outcomes, produce fewer higher-order corneal aberrations and decrease rejection rates. However, donor preparation, increased intra-operative times, and problems with donor attachment in DMEK are all important limitations.

There are three potential mechanisms by which DMEK may provide better visual acuity outcomes than DSAEK; graft thickness, interface haze and corneal higher-order aberrations. Graft thickness has been correlated with best spectacle corrected visual acuity (BSCVA) outcomes among thinner grafts. One retrospective case series found that 71% of thin endothelial grafts (defined as <131μm) had BSCVA of 20/25 or better while only 50% of thick grafts (defined as ≥131) achieved this. In addition, higher-order aberrations, in particular of the posterior cornea, are increased after DSAEK. Theoretically, given the decreased tissue transplanted after DMEK this would be lessened, however, one retrospective series looking at higher order aberrations in DMEK compared with DSAEK found no difference in posterior aberrations of the central 4.0 mm zone between the two groups. Finally, interface haze may be increased in DSAEK and has been correlated with BSCVA.

Ultrathin DSAEK involves donor preparation with a deep microkeratome pass to produce donor grafts less than 100 um thick. This procedure may have similar results to DMEK but without the technical difficulties. Several large prospective series show similar visual outcome results and rates of immunologic rejection between ultrathin DSAEK and DMEK, however comparisons are difficult. This comparative effectiveness clinical trial could directly address these important issues. The investigators also anticipate that secondary analyses of the trial data will allow us to address several more.

ELIGIBILITY:
Inclusion Criteria:

* Damaged or diseased endothelium from Fuchs or Pseudophakic Bullous Keratopathy
* Good candidates for corneal transplantation for either DMEK or DSAEK
* Willingness and ability to undergo a cornea transplantation
* Willingness to participate in follow-up visits

Exclusion Criteria:

* Participants who are decisionally and/or cognitively impaired
* Participants who are not suitable for the DMEK or DSAEK surgeries
* Prior Endothelial Keratoplasty (EK) or any other ophthalmic surgery except uncomplicated cataract surgery
* Indication for surgery that is not suitable for EK (e.g. keratoconus, stromal dystrophies and scars)
* Presence of a condition that increases the probability for failure (e.g., heavily vascularized cornea, uncontrolled uveitis)
* Other primary endothelial dysfunction conditions including posterior polymorphous corneal dystrophy and congenital hereditary corneal dystrophy
* Aphakia, or anterior chamber intraocular lens (IOL) in study eye prior to or anticipated during EK
* Planned intraocular lens exchange of an anterior chamber IOL with a posterior chamber IOL in study at time of study EK
* Pre-operative central sub-epithelial or stromal scarring that the investigator believes is visually significant and could impact post-operative stromal clarity assessment
* Peripheral anterior synechiae (iris to angle) in the angle greater than a total of three clock hours
* Hypotony (Intraocular pressure <10mmHg)
* Uncontrolled (defined as intraocular pressure >25mmHg) glaucoma Visually significant optic nerve or macular pathology
* Visually significant optic nerve or macular pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-01-22 (Actual); Primary Completion 2018-04-04 (Actual); Study Completion 2023-05-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Winston Chamberlain, MD, PhD, Principal Investigator — Oregon Health and Science University; Jennifer Rose-Nussbaumer, MD, Principal Investigator — University of California, San Francisco; Charles Lin, MD, Principal Investigator — Stanford University
Locations (3):
- United States (3):
  - Byers Eye Institute, Stanford University, Palo Alto, California
  - F. I. Proctor Foundation, University of California, San Francisco, San Francisco, California
  - Casey Eye Institute, Oregon Health & Science University, Portland, Oregon

REFERENCES:
- [Background] Price FW Jr, Price MO. Evolution of endothelial keratoplasty. Cornea. 2013 Nov;32 Suppl 1:S28-32. doi: 10.1097/ICO.0b013e3182a0a307. PMID 24104929
- [Background] Chen ES, Terry MA, Shamie N, Hoar KL, Friend DJ. Descemet-stripping automated endothelial keratoplasty: six-month results in a prospective study of 100 eyes. Cornea. 2008 Jun;27(5):514-20. doi: 10.1097/ICO.0b013e3181611c50. PMID 18520497
- [Background] Ham L, Dapena I, van Luijk C, van der Wees J, Melles GR. Descemet membrane endothelial keratoplasty (DMEK) for Fuchs endothelial dystrophy: review of the first 50 consecutive cases. Eye (Lond). 2009 Oct;23(10):1990-8. doi: 10.1038/eye.2008.393. Epub 2009 Jan 30. PMID 19182768
- [Background] Dirisamer M, van Dijk K, Dapena I, Ham L, Oganes O, Frank LE, Melles GR. Prevention and management of graft detachment in descemet membrane endothelial keratoplasty. Arch Ophthalmol. 2012 Mar;130(3):280-91. doi: 10.1001/archophthalmol.2011.343. Epub 2011 Nov 14. PMID 22084160
- [Background] Kruse FE, Laaser K, Cursiefen C, Heindl LM, Schlotzer-Schrehardt U, Riss S, Bachmann BO. A stepwise approach to donor preparation and insertion increases safety and outcome of Descemet membrane endothelial keratoplasty. Cornea. 2011 May;30(5):580-7. doi: 10.1097/ico.0b013e3182000e2e. PMID 21598430
- [Background] Rudolph M, Laaser K, Bachmann BO, Cursiefen C, Epstein D, Kruse FE. Corneal higher-order aberrations after Descemet's membrane endothelial keratoplasty. Ophthalmology. 2012 Mar;119(3):528-35. doi: 10.1016/j.ophtha.2011.08.034. Epub 2011 Dec 22. PMID 22197439
- [Background] Busin M, Madi S, Santorum P, Scorcia V, Beltz J. Ultrathin descemet's stripping automated endothelial keratoplasty with the microkeratome double-pass technique: two-year outcomes. Ophthalmology. 2013 Jun;120(6):1186-94. doi: 10.1016/j.ophtha.2012.11.030. Epub 2013 Mar 1. PMID 23466268
- [Background] Guerra FP, Anshu A, Price MO, Giebel AW, Price FW. Descemet's membrane endothelial keratoplasty: prospective study of 1-year visual outcomes, graft survival, and endothelial cell loss. Ophthalmology. 2011 Dec;118(12):2368-73. doi: 10.1016/j.ophtha.2011.06.002. Epub 2011 Aug 27. PMID 21872938
- [Derived] Ang MJ, Chamberlain W, Lin CC, Pickel J, Austin A, Rose-Nussbaumer J. Effect of Unilateral Endothelial Keratoplasty on Vision-Related Quality-of-Life Outcomes in the Descemet Endothelial Thickness Comparison Trial (DETECT): A Secondary Analysis of a Randomized Clinical Trial. JAMA Ophthalmol. 2019 Jul 1;137(7):747-754. doi: 10.1001/jamaophthalmol.2019.0877. PMID 31046075
- [Derived] Chamberlain W, Lin CC, Austin A, Schubach N, Clover J, McLeod SD, Porco TC, Lietman TM, Rose-Nussbaumer J. Descemet Endothelial Thickness Comparison Trial: A Randomized Trial Comparing Ultrathin Descemet Stripping Automated Endothelial Keratoplasty with Descemet Membrane Endothelial Keratoplasty. Ophthalmology. 2019 Jan;126(1):19-26. doi: 10.1016/j.ophtha.2018.05.019. Epub 2018 Jun 23. PMID 29945801

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: eyes
Groups:
- UT-DSAEK: Type of corneal transplant; Tissue grafts will be cut to the right thickness using a microkeratome prepared at the eye bank per standard eye bank protocol (about 60-90 microns thick). A 4 mm corneal incision will be used, with Endoserter as the means of inserting the graft, an FDA approved device for this purpose.
  UT-DSAEK
  Endoserter: The Endoserter, a corneal endothelium device, is an approved FDA device. This will be used to insert and position the graft into the anterior chamber during endothelial replacement surgery. It is a sterile, single-use instrument.
  Prednisolone: Prednisolone is a corticosteroid used to alleviate swelling post-surgery.
  Ofloxacin: Ofloxacin is an antibiotic used to treat bacterial infections of the eye.
  Tropicamide: Tropicamide is a prescription drug used to dilate pupils during an eye exam.
  Phenylephrine: Phenylephrine is a prescription drug used to dilate pupils during an eye exam.
- DMEK: Type of corneal transplant; Endothelial grafts will be pre-peeled at the eyebank (70%). In the operating room the remaining 30% will be peeled, and the endothelium will be stained with trypan blue. A 3.5 mm corneal incision will be used and the graft will be inserted with a modified jones tube injector. The tap technique will be used to position the graft.
  DMEK
  Prednisolone: Prednisolone is a corticosteroid used to alleviate swelling post-surgery.
  Ofloxacin: Ofloxacin is an antibiotic used to treat bacterial infections of the eye.
  Tropicamide: Tropicamide is a prescription drug used to dilate pupils during an eye exam.
  Phenylephrine: Phenylephrine is a prescription drug used to dilate pupils during an eye exam.
  Jones Tube: The Jones Tube will be used to insert the graft into a 3.5 mm corneal incision during endothelial replacement surgery.
Period: Overall Study
Arm/Group | UT-DSAEK | DMEK
Started | 19; 25 eyes | 19; 25 eyes
3-Month Follow-Up | 19; 25 eyes | 19; 25 eyes
6-Month Follow-Up | 19; 25 eyes | 18; 24 eyes
12-Month Follow-Up | 19; 25 eyes | 19; 25 eyes
Completed | 18; 24 eyes | 18; 23 eyes
Not Completed | 1; 1 eyes | 1; 2 eyes

BASELINE CHARACTERISTICS:
Units Other Than Participants: eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | UT-DSAEK | DMEK | Total
Number analyzed (Participants) | 19 | 19 | 38
Number analyzed (eyes) | 25 | 25 | 50
Age, Continuous [Mean (Full Range); unit: years] | 68 [51 to 95] | 68 [61 to 81] | 68 [51 to 95]
Sex: Female, Male [Count of Units; unit: eyes]
  Female | 16 | 13 | 29
  Male | 9 | 12 | 21
Race (NIH/OMB) [Count of Units; unit: eyes]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 24 | 24 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: eyes]
  United States | 25 | 25 | 50
Diagnosis [Count of Units; unit: eyes]
  Fuch's Dystrophy | 24 | 24 | 48
  Pseudophakic Bullous Keratopathy | 1 | 1 | 2
Best Spectacle-Corrected Visual Acuity (logMAR) [Mean (Standard Deviation); unit: logMAR] — ETDRS Best spectacle-corrected visual acuity in logarithm of the minimum angle of resolution (logMAR) units
  logMAR | 0.27 (0.21) | 0.34 (0.29) | 0.30 (0.25)
Surgery [Count of Units; unit: eyes]
  Pseudophakic Endothelial Keratoplasty | 8 | 7 | 15
  Triple Endothelial Keratoplasty | 17 | 18 | 35
Donor Age [Mean (Full Range); unit: years] | 64 [54 to 75] | 62 [50 to 76] | 63 [50 to 76]
Donor Sex [Count of Units; unit: eyes]
  Female | 8 | 5 | 13
  Male | 17 | 20 | 37
Donor Death to Preservation Time [Mean (Standard Deviation); unit: hours] | 9 (4) | 9 (3) | 9 (4)
Donor Death to Surgery Time [Mean (Standard Deviation); unit: days] | 6 (1) | 6 (1) | 6 (1)
Donor Endothelial Cell Count (pre-processing) [Mean (Standard Deviation); unit: cells/mm^2] | 2792 (210) | 2797 (222) | 2795 (214)
Donor Endothelial Cell Count (post-processing) [Mean (Standard Deviation); unit: cells/mm^2] | 2796 (238) | 2771 (150) | 2783 (197)
Donor Central Graft Thickness (UT-DSAEK only) [Mean (Full Range); unit: mm] | 73 [37 to 88] | NA [NA to NA] — N/A to DMEK grafts | 73 [37 to 88]
Central Corneal Thickness [Mean (Standard Deviation); unit: microns] — Population: missing one value
  microns
    number analyzed (Participants) | 18 | 19 | 37
    number analyzed (eyes) | 24 | 25 | 49
    (all) | 610 (44) | 608 (52) | 609 (48)
Spherical Equivalent [Mean (Standard Deviation); unit: diopters] | -0.4 (1.9) | -0.8 (2.2) | -0.6 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: Best Spectacle-Corrected Visual Acuity
Description: The BSCVA was recorded at 4 meters by a masked refractionist certified for the study using a protocol adapted from the Age-Related Eye Disease Study using Early Treatment Diabetic Retinopathy Study charts: chart R(2110), chart 1(2111), and chart 2(2112) (Precision Vision, Woodstock, IL).
Time Frame: 6 months
Population: One patient lost to followup
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | UT-DSAEK | DMEK
Number analyzed (Participants) | 19 | 18
Number analyzed (eyes) | 25 | 24
logMAR | 0.22 (0.16) | 0.05 (0.11)
Statistical Analysis 1: Comparison: UT-DSAEK vs DMEK; Test type: Superiority; p < 0.001, Regression, Linear; Multiple linear regression model with a covariate for baseline visual acuity; Coefficient = -1.8, 95% CI 2-sided [-2.8 to -1.0] — Coefficient reported in lines, comparing DMEK to UT-DSAEK. Compared to UT-DSAEK, DMEK had 1.8 lines better vision at 6 months

2. Secondary Outcome: Best Spectacle-Corrected Visual Acuity
Description: as for outcome 1
Time Frame: 3 and 12 months
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | UT-DSAEK | DMEK
Number analyzed (Participants) | 19 | 19
Number analyzed (eyes) | 25 | 25
logMAR
  3 Months | 0.24 (0.21) | 0.11 (0.13)
  12 Months | 0.16 (0.18) | 0.04 (0.12)
Statistical Analysis 1: Comparison: UT-DSAEK vs DMEK; Comparison of 3-Month Visual Acuity Between Groups; Test type: Superiority; p = 0.002, Regression, Linear; Multiple linear regression model with a covariate for baseline visual acuity; Coefficient = -1.5, 95% CI 2-sided [-2.5 to -0.6] — Coefficient reported in lines, comparing DMEK to UT-DSAEK. Compared to UT-DSAEK, DMEK had 1.5 lines better vision at 3 months
Statistical Analysis 2: Comparison: UT-DSAEK vs DMEK; Comparison of 12 Month Visual Acuity Between Groups; Test type: Superiority; p < 0.001, Regression, Linear; Multiple linear regression model with a covariate for baseline visual acuity; Coefficient = -1.4, 95% CI 2-sided [-2.2 to -0.7] — Coefficient reported in lines, comparing DMEK to UT-DSAEK. Compared to UT-DSAEK, DMEK had 1.4 lines better vision at 12 months

3. Secondary Outcome: Best Spectacle-Corrected Visual Acuity
Description: as for outcome 1
Time Frame: 24 Months
Measure: Mean (Standard Deviation); unit: LogMar
Units Other Than Participants: eyes
Arm/Group | UT-DSAEK | DMEK
Number analyzed (Participants) | 19 | 19
Number analyzed (eyes) | 25 | 25
LogMar | 0.15 (0.15) | 0.09 (0.16)

4. Secondary Outcome: Endothelial Cell Count
Time Frame: 3, 6, 12 months
Measure: Mean (Standard Deviation); unit: cells/mm^2
Units Other Than Participants: eyes
Arm/Group | UT-DSAEK | DMEK
Number analyzed (Participants) | 19 | 19
Number analyzed (eyes) | 25 | 25
cells/mm^2
  3 Months | 2114 (357) | 2037 (495)
  6 Months | 2113 (301) | 1963 (425)
  12 Months | 2070 (292) | 1855 (448)
Statistical Analysis 1: Comparison: UT-DSAEK vs DMEK; Test type: Superiority; p = 0.53, t-test, 2 sided; Coefficient = -77, 95% CI 2-sided [-326 to 172] — Comparing DMEK to UT-DSAEK at 3 months
Statistical Analysis 2: Comparison: UT-DSAEK vs DMEK; Test type: Superiority; p = 0.17, t-test, 2 sided; Coefficient = -150, 95% CI 2-sided [-356 to 66] — Comparing DMEK to UT-DSAEK at 6 months
Statistical Analysis 3: Comparison: UT-DSAEK vs DMEK; Test type: Superiority; p = 0.051, t-test, 2 sided; Coefficient = -215, 95% CI 2-sided [-430 to -0.4] — Comparing DMEK to UT-DSAEK at 12 months

5. Secondary Outcome: Endothelial Cell Count
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: cells/mm^2
Units Other Than Participants: eyes
Arm/Group | UT-DSAEK | DMEK
Number analyzed (Participants) | 19 | 19
Number analyzed (eyes) | 25 | 25
cells/mm^2 | 1626 (362) | 1400 (498)

6. Secondary Outcome: Corneal Higher-Order Aberrations
Description: Corneal anterior and posterior surface higher-order aberrations (HOA) were measured with Scheimpflug imaging (Pentacam) before surgery and at 3, 6, and 12 months post-operatively. Zernike orders 3-8 were calculated at 4.0- and 6.0-mm-diameter optical zones. The results reported here represent total HOA (Sum of Zernike orders 3-8). Note a single observation was not available for one eye in the DMEK group at 6 months, this was analyzed with last observation carried forward.
Time Frame: 3, 6, 12 months
Measure: Mean (Standard Deviation); unit: root mean square in micrometers
Units Other Than Participants: eyes
Arm/Group | UT-DSAEK | DMEK
Number analyzed (Participants) | 19 | 19
Number analyzed (eyes) | 25 | 25
root mean square in micrometers
  3 Months Anterior Cornea 4.0-mm | 0.274 (0.223) | 0.288 (0.104)
  3 Months Posterior Cornea 4.0-mm | 0.217 (0.110) | 0.116 (0.056)
  3 Months Anterior Cornea 6.0-mm | 0.897 (0.800) | 0.829 (0.367)
  3 Months Posterior Cornea 6.0-mm | 0.621 (0.308) | 0.346 (0.153)
  6 Months Anterior Cornea 4.0-mm | 0.230 (0.110) | 0.243 (0.100)
  6 Months Posterior Cornea 4.0-mm | 0.179 (0.067) | 0.095 (0.031)
  6 Months Anterior Cornea 6.0-mm | 0.739 (0.371) | 0.724 (0.337)
  6 Months Posterior Cornea 6.0-mm | 0.505 (0.217) | 0.288 (0.089)
  12 Months Anterior Cornea 4.0-mm | 0.228 (0.108) | 0.241 (0.100)
  12 Months Posterior Cornea 4.0-mm | 0.159 (0.068) | 0.098 (0.028)
  12 Months Anterior Cornea 6.0-mm | 0.725 (0.344) | 0.723 (0.328)
  12 Months Posterior Cornea 6.0-mm | 0.459 (0.206) | 0.284 (0.073)

7. Secondary Outcome: Corneal Higher-Order Aberrations
Description: As measured by Pentacam
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: root mean square in micrometers
Units Other Than Participants: eyes
Groups:
- DSAEK: Type of corneal transplant; Tissue grafts will be cut to the right thickness using a microkeratome prepared at the eye bank per standard eye bank protocol (about 60-90 microns thick). A 4 mm corneal incision will be used, with Endoserter as the means of inserting the graft, an FDA approved device for this purpose.
  DSAEK
  Endoserter: The Endoserter, a corneal endothelium device, is an approved FDA device. This will be used to insert and position the graft into the anterior chamber during endothelial replacement surgery. It is a sterile, single-use instrument.
  Prednisolone: Prednisolone is a corticosteroid used to alleviate swelling post-surgery.
  Ofloxacin: Ofloxacin is an antibiotic used to treat bacterial infections of the eye.
  Tropicamide: Tropicamide is a prescription drug used to dilate pupils during an eye exam.
  Phenylephrine: Phenylephrine is a prescription drug used to dilate pupils during an eye exam.
Arm/Group | DSAEK | DMEK
Number analyzed (Participants) | 19 | 19
Number analyzed (eyes) | 25 | 25
root mean square in micrometers
  24 Months Anterior Cornea 4.0-mm | 0.215 (0.136) | 0.211 (0.008)
  24 Months Posterior Cornea 4.0-mm | 0.155 (0.075) | 0.086 (0.029)
  24 Months Anterior Cornea 6.0-mm | 0.707 (0.389) | 0.679 (0.314)
  24 Months Posterior Cornea 6.0-mm | 0.450 (0.216) | 0.260 (0.008)

8. Secondary Outcome: Interface Haze
Description: As measured by Pentacam densitometry
Time Frame: 3, 6, 12 months
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | UT-DSAEK | DMEK
Number analyzed (Participants) | 19 | 19
Number analyzed (eyes) | 25 | 25
eyes
  Mild Interface Haze at 3 months | 2 | 1
  Moderate Interface Haze at 3 months | 0 | 0
  Severe Interface Haze at 3 months | 0 | 0
  Mild Interface Haze at 6 months | 2 | 1
  oderate Interface Haze at 6 months | 1 | 0
  Severe Interface Haze at 6 months | 0 | 0
  Mild Interface Haze at 12 months | 0 | 0
  oderate Interface Haze at 12 months | 0 | 0
  Severe Interface Haze at 12 months | 0 | 0

9. Secondary Outcome: Interface Haze
Description: As measured by Pentacam densitometry
Time Frame: 24 months
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | UT-DSAEK | DMEK
Number analyzed (Participants) | 19 | 19
Number analyzed (eyes) | 25 | 25
eyes
  Mild Interface Haze at 24 months | 0 | 0
  Moderate Interface Haze at 24 months | 1 | 0
  Severe Interface Haze at 24 months | 0 | 0

10. Secondary Outcome: National Eye Institute - Visual Functioning Questionnaire (NEI-VFQ)
Description: The National Eye Institute has developed the validated Visual Functioning Questionnaire (NEI-VFQ) to assess the effect of ocular conditions and vision on patient quality of life. The answers to the questionnaire are transformed into sub-scales, including: general health, general vision, ocular pain, near activities, distance activities, social functioning, mental health, role difficulties, dependency, driving, color vision, peripheral vision. Participants are assigned a numerical value for each sub-scale based on their answers between 0-100, where higher numbers indicate better visual function. These sub-scales are then combined according to National Eye Institute guidelines into an overall composite score for each participant. This overall composite score is also on a scale of 0-100, where higher numbers indicate better visual function.
  Composite score based on National Eye Institute guidelines.
Time Frame: Baseline, 12 months
Population: For this analysis, all "second eyes" (enrolled eyes belonging to a patient that had enrolled their other eye and already had surgery on that eye as part of this study) were removed. For this reason the total number of eyes equals the total number of participants.
Measure: Mean (Standard Deviation); unit: Composite scores on a scale
Units Other Than Participants: eyes
Arm/Group | UT-DSAEK | DMEK
Number analyzed (Participants) | 19 | 19
Number analyzed (eyes) | 19 | 19
Composite scores on a scale
  Baseline | 72.5 (13.4) | 72.3 (15.2)
  12 Months: number analyzed (Participants) | 14 | 12
  12 Months: number analyzed (eyes) | 14 | 12
  12 Months | 85.9 (9.1) | 87.3 (9.5)
Statistical Analysis 1: Comparison: UT-DSAEK vs DMEK; Test type: Superiority; p = 0.70, t-test, 2 sided

11. Secondary Outcome: Graft Failure/Graft Rejection
Time Frame: Baseline 12 months
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | UT-DSAEK | DMEK
Number analyzed (Participants) | 19 | 19
Number analyzed (eyes) | 25 | 25
eyes
  Graft Rejection | 0 | 0
  Graft Failure | 1 | 1

12. Secondary Outcome: Graft Failure/Graft Rejection
Time Frame: Baseline to 24 months
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | DSAEK | DMEK
Number analyzed (Participants) | 19 | 19
Number analyzed (eyes) | 25 | 25
eyes
  Graft Rejection | 0 | 0
  Graft Failure | 1 | 1
  Eyes with No Graft Failure or Rejection | 24 | 24

13. Other Pre Specified Outcome: Refraction
Description: Manifest refraction using phoropter
Time Frame: 3, 6, 12, 24 months
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Graft Thickness
Description: As measured by Optical coherence tomography (OCT) and Pachymetry
Time Frame: 3, 6, 12, 24 months
Measure: Mean (95% Confidence Interval); unit: root mean square in micrometers
Units Other Than Participants: eyes
Arm/Group | UT-DSAEK | DMEK
Number analyzed (Participants) | 19 | 19
Number analyzed (eyes) | 25 | 25
root mean square in micrometers
  3 months | 589.36 [568.40 to 614.50] | 516.5 [499.40 to 533.35]
  6 months | 592.24 [573.92 to 612.84] | 519.67 [504.75 to 533.88]
  12 months | 585.96 [569.32 to 603.12] | 521.36 [506.28 to 536.32]
  24 months | 593.67 [577.08 to 612.21] | 526.88 [512.20 to 541.28]

15. Other Pre Specified Outcome: Operative Times
Time Frame: Baseline
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Adverse Events/Complication Rates
Description: composite measure
Time Frame: 3, 6, 12, 24 months
Measure: Number; unit: new adverse events reported
Units Other Than Participants: eyes
Arm/Group | UT-DSAEK | DMEK
Number analyzed (Participants) | 19 | 19
Number analyzed (eyes) | 25 | 25
new adverse events reported
  Adverse Events at 3 months | 4 | 6
  Adverse Events at 6 months | 4 | 5
  Adverse Events at 12 months | 1 | 4
  Adverse Events at 24 months | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 months
Description: Adverse events are reported by eye (N = 50), not by participant (N = 38).
Arm/Group | UT-DSAEK | DMEK
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 9/25 | 7/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UT-DSAEK (N=25) | DMEK (N=25)
Glaucoma (nonsurgical) (Eye disorders) | 2 | 2
Glaucoma (surgical) (Eye disorders) | 1 | 1
Graft displacement (Eye disorders) | 1 | 0
Graft failure (Eye disorders) | 1 | 1
Graft rejection (Eye disorders) | 0 | 0
Infectious keratitis (Eye disorders) | 0 | 0
Posterior synechiae (Eye disorders) | 0 | 1
Re-bubble (Eye disorders) | 1 | 6
Retinal tear (Eye disorders) | 0 | 1
Visually significant central epithelial opacity (Eye disorders) | 1 | 0
Intralocular lens repositioning (Eye disorders) | 0 | 1
Epiretinal membrane and lamellar hole (Eye disorders) | 0 | 1
Cystoid macular edema (Eye disorders) | 0 | 1
Visual disturbance (Eye disorders) | 1 | 1
Postoperative day 1 pupillary block (Eye disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-10-02): https://cdn.clinicaltrials.gov/large-docs/37/NCT02373137/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-07): https://cdn.clinicaltrials.gov/large-docs/37/NCT02373137/SAP_001.pdf